CLINICAL TRIAL: NCT00731510
Title: MEDEX Hidden Valley 2008
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Expeditions Ltd (Other)
Collaborators: Bangor University (Other); Science in Sport (Unknown); Plans Branch of Headquarters Army Recruiting and Training Division (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 08/WNo01/16
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Hypoxia
Keywords: Acute mountain sickness; Body composition,Hypoxia; Carbohydrate supplementation; Expedition,; Hydration,; Hypoxia; Performance
MeSH Terms: conditions — Hypoxia; Altitude Sickness | interventions — Aspartame

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Carbohydrate supplements (drinks and gels)
  Interventions: Dietary Supplement: Carbohydrate energy drink
- 2 (Placebo Comparator): Primarily Aspartame plus natural flavourings. Powder dissolved in water to provide non-distinguishable placebo drink.
  Interventions: Dietary Supplement: Aspartame

INTERVENTIONS:
Dietary Supplement: Carbohydrate energy drink — Complex carbohydrates including maltodextrin (97%) dissolved in water to make a a 10% solution, or dissolved in 25mL gels. Ad libitum. Twenty two days.
  Other Names: PSP22 Energy, Science in Sport, Blackburn, UK
  Arms: 1
Dietary Supplement: Aspartame — Aspartame dissolved in water, ad libitum, 22 days.
  Other Names: Science in Sport, Blackburn, UK
  Arms: 2

SUMMARY:
During a multi-week expedition to the Himalaya, we aim to investigate i) whether dietary supplementation with carbohydrate drinks and gels can improve physical performance; and ii) the underlying mechanisms for any observed changes in performance.

We hypothesise that i) carbohydrate supplementation will improve physical performance; and ii) the underlying mechanism of this improvement in performance will include maintenance of body glycogen (sugar) stores, prevention of dehydration and decrease in the incidence of acute mountain sickness.

ELIGIBILITY:
Inclusion Criteria:

* a healthy enthusiasm for the outdoors and/or a passion for research in remote and difficult circumstances

Exclusion Criteria:

* Persons with Phenylketonuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Performance (time to complete a physical performance task) | Mid study

SECONDARY OUTCOMES:
Body composition | Pre, mid and post study
Hydration status | Pre, mid and post study
Body glucose stores | Pre, mid and post study
Oxygen delivery | Pre, mid and post study
Acute mountain sickness | Every day
Spontaneous physical activity level | Pre, mid and post study
Rating of perceived exertion during a stepping task | Pre, mid and post study

CONTACTS AND LOCATIONS:
Overall Officials: Jamie H Macdonald, PhD, Principal Investigator — Bangor University; Samuel J Oliver, PhD, Principal Investigator — Bangor University
Locations (1):
- Medical Expeditions Ltd, Pinfold, Hyssington, Montgomery, Powys, United Kingdom

REFERENCES:
- [Derived] Macdonald JH, Oliver SJ, Hillyer K, Sanders S, Smith Z, Williams C, Yates D, Ginnever H, Scanlon E, Roberts E, Murphy D, Lawley J, Chichester E. Body composition at high altitude: a randomized placebo-controlled trial of dietary carbohydrate supplementation. Am J Clin Nutr. 2009 Nov;90(5):1193-202. doi: 10.3945/ajcn.2009.28075. Epub 2009 Sep 30. PMID 19793859